CLINICAL TRIAL: NCT03927469
Title: Analysis Of The Patients Who Need Rehospitalization Due To Stroke Rehabilitation Only
Acronym: RSR
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tuğba Aydın, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: IstPMRTRH-449
Record Dates: First submitted 2019-03-20; First posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Stroke Rehabilitation
MeSH Terms: interventions — Aging; Sex; Seasons; CAF protocol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospitalisation group: The patients who were hospitalized in the hospital between January 2015 and July 2018, according to ICD 10 code; hemiplegia (G81), flaccid hemiplegia (G81.0), hemiplegia, unspecified (G81.9), Spastic hemiplegia (G81.1) scanned from the hospital database.
  Interventions: Other: age, sex, hemiplegic side, stroke duration, First hospitalisation duration (day)
- Re-hospitalisation group.: The patients who were re-hospitalized in the hospital between January 2015 and July 2018, according to ICD 10 code; hemiplegia (G81), flaccid hemiplegia (G81.0), hemiplegia, unspecified (G81.9), Spastic hemiplegia (G81.1) scanned from the hospital database.
  Interventions: Other: age, sex, hemiplegic side, stroke duration, First hospitalisation duration (day)

INTERVENTIONS:
Other: age, sex, hemiplegic side, stroke duration, First hospitalisation duration (day) — This is a retrospiective descriptive study
  Other Names: Corelation of data, FAC: Functional Ambulation Classification and age, stroke duration, Season, stroke Etiology, Brunnstrom, FAC

SUMMARY:
The aim of this study was to investigate the clinical and laboratory data of patients who were rehospitalised due to "stroke rehabilitation cause only" The patients who were hospitalized in the hospital between January 2015 and July 2018, according to ICD 10 code; hemiplegia (G81), flaccid hemiplegia (G81.0), hemiplegia, unspecified (G81.9), Spastic hemiplegia (G81.1) scanned from the hospital database.

DETAILED DESCRIPTION:
All comorbid diseases were included to rehospitalisation rates in stroke patients in the literature. The aim of this study was to investigate the clinical and laboratory data of patients who were rehospitalised due to "stroke rehabilitation cause only" The patients who were hospitalized in the hospital between January 2015 and July 2018, according to ICD 10 code; hemiplegia (G81), flaccid hemiplegia (G81.0), hemiplegia, unspecified (G81.9), Spastic hemiplegia (G81.1) scanned from the hospital database.

There were 554 patients with these diagnoses. 9 patients of them were excluded because of the hemiplegic due to trauma, cancer and intracranial operation. Detailed epicrisis of 545 patients with ischemic or hemorrhagic stroke were examined. 328 patients who did not have missing data were included in the study. Age, sex, hemiplegia etiology, admission season, hemiplegia time, hemiplegic side, 25 (OH) vitamin D and vitamin B12 levels, brunnstrom stage of upper extremity, lower extremity and hand Functional Ambulation Classification (FAC).

Brunnstrom staging was used to identify motor function with 6 levels in the upper extremity and hand. ROM for abduction, flexion, internal rotation, and external rotation were passively measured. Brunnstrom staging was used to evaluate motor development, and stroke patients were defined as 6 stages. The flask phase without the lowest voluntary movement is considered to be stage 1, while the presence of isolated movements is considered to be stage 6. In the Brunstromm staging, upper, lower extremity and hand evaluation are performed separately.

FAC is defined as 5 stages according to the basic motor skills required for functional ambulation. FAC stage 0 is used for non-functional ambulation, stage 5 is used for independent walking at each speed and ground.

ELIGIBILITY:
Inclusion Criteria:

* Being hospitalized in the hospital between January 2015 and July 2018, according to ICD 10 code; hemiplegia (G81), flaccid hemiplegia (G81.0), hemiplegia, unspecified (G81.9), Spastic hemiplegia (G81.1)
* Being ischemic or hemorrhagic stroke

Exclusion Criteria:

* Being hemiplegic due to trauma, cancer and intracranial operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who were hospitalized in the hospital between January 2015 and July 2018, according to ICD 10 code; hemiplegia (G81), flaccid hemiplegia (G81.0), hemiplegia, unspecified (G81.9), Spastic hemiplegia (G81.1) were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Rehospitalisation rates | 3 YEARS
  rehospitalisation rates. Data will given as percent

SECONDARY OUTCOMES:
Serum vitamin D level | 3 YEARS
  Serum 25 (OH) vitamin D level. Unit of this parameter is U/L
Serum vitamin B12 level | 3 YEARS
  Serum B12 level. Unit of this parameter is U/L

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA AYDIN, Study Chair — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ottenbacher KJ, Graham JE, Ottenbacher AJ, Lee J, Al Snih S, Karmarkar A, Reistetter T, Ostir GV. Hospital readmission in persons with stroke following postacute inpatient rehabilitation. J Gerontol A Biol Sci Med Sci. 2012 Aug;67(8):875-81. doi: 10.1093/gerona/glr247. Epub 2012 Mar 2. PMID 22389457
- [Background] Sun Y, Lee SH, Heng BH, Chin VS. 5-year survival and rehospitalization due to stroke recurrence among patients with hemorrhagic or ischemic strokes in Singapore. BMC Neurol. 2013 Oct 3;13:133. doi: 10.1186/1471-2377-13-133. PMID 24088308